CLINICAL TRIAL: NCT03900897
Title: Expanded Indications in the MED-EL Pediatric Cochlear Implant Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G180269; NCT04130113 (obsolete NCT alias)
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Cochlear Implants

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, non-randomized, repeated-measures design with two study arms as follows. Prospective: interventional study arm with prospective enrollment and treatment through one year of implant use. Retrospective: observational study arm with retrospective protocol for systematic chart review of patients with at least one year of implant use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Prospective (Experimental): Detailed interventions and outcome measures refer to the prospective, experimental study arm. The prospective arm is active but not enrolling.
  Interventions: Device: MED-EL SYNCHRONY PIN Cochlear Implant
- Retrospective (Other): Study identification, sponsor/collaborators, oversight, purpose, indications, and primary endpoints for the retrospective, observational study arm align with the prospective study arm. The retrospective arm will be enrolling by invitation for chart review of subjects implanted with a MED-EL cochlear implant under 6 years of age between January 2005 and October 2020. The specific devices and outcome measures will vary slightly for retrospective subjects, based on what was clinically available and used at the time of implantation.
  Interventions: Other: Cochlear Implant

INTERVENTIONS:
Device: MED-EL SYNCHRONY PIN Cochlear Implant — Subjects will be implanted with the MED-EL SYNCHRONY PIN Cochlear Implant System with +FLEX24, +FLEX28, +FLEXSOFT electrode arrays. Subjects will be fit with the SONNETEAS (ear-level) and/or RONDO 2 (single-unit) external audio processors.
  Other Names: SYNCHRONY +FLEXSOFT; SYNCHRONY +FLEX28; SYNCHRONY +FLEX24
  Arms: Prospective
Other: Cochlear Implant — Chart review of subjects implanted with a MED-EL cochlear implant under 6 years of age between January 2005 and October 2020.
  Arms: Retrospective

SUMMARY:
The purpose of this investigation is to demonstrate the safety and effectiveness of MED-EL cochlear implants in children 7 months to 5 years, 11 months of age who fall outside the current FDA-approved candidacy criteria and, yet, continue to demonstrate insufficient functional access to sound with appropriately fit hearing aids and aural habilitation.

ELIGIBILITY:
Inclusion Criteria:

* Children 7 months to 5 years 11 months of age at the time of implantation
* Bilateral, severe to profound sensorineural hearing loss (SNHL) in the high frequencies and

  * For subjects implanted under 12 months of age: bilateral, severe to profound SNHL in the low frequencies
  * For subjects implanted at 12 months to 5 years 11 months of age: bilateral, mild to profound sensorineural hearing loss in the low frequencies
* Insufficient functional access to sound with appropriately fit amplification and aural habilitation
* Objective measures consistent with repeatable unaided audiometric thresholds for subjects under 12 months of age
* Radiologic evidence of potential for full insertion with one of the included electrode arrays
* Ability to undergo general anesthesia
* At least one parent/guardian who is fluent in one of the available languages of the LEAQ
* Parental commitment to study parameters

Exclusion Criteria:

* Magnetic Resonance Imaging (MRI) evidence of cochlear nerve deficiency
* Active middle ear infection
* Permanent conductive hearing loss
* Treatable mixed hearing loss
* Current or history of meningitis
* Common cavity
* Skin or scalp condition precluding use of external audio processor
* Suspected cognitive impairment, organic brain dysfunction, or syndromic etiology that may affect performance
* ASA (American Society of Anesthesiologists) Class 3 or higher in subjects under 12 months of age
* History of prior use of a hearing implant
* Unrealistic parental/patient expectations
* Child is not able to complete speech perception testing in English

Ages: 7 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 247 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Total Score on LittlEARS Auditory Questionnaire (LEAQ) | Up to 12 Months Post-Activation
  Clinical success defined as a Total Score of 25 or more on the LittLEARS Auditory Questionnaire (LEAQ). Total Score ranges from zero to 35, with higher scores indicating development of increasingly complex listening skills.
Percent correct on Multisyllabic Lexical Neighborhood Test (MLNT)/Lexical Neighborhood Test (LNT) | Up to 12 Months Post-Activation
  Clinical success defined as an improvement of 10 percentage points or more on MLNT/LNT.
Number and proportion of subjects experiencing device- and/or procedure-related adverse events. | Up to 12 Months Post-Activation
  Adverse events will be collected and reported throughout the duration of the study.

SECONDARY OUTCOMES:
Total Score on LittlEARS Auditory Questionnaire (LEAQ) | Up to 12 Months Post-Activation
  Change from baseline in Total Score on the LittlEARS Auditory Questionnaire (LEAQ). Total Score ranges from zero to 35, with higher scores indicating development of increasingly complex listening skills. The LittlEARS Auditory Questionnaire is intended for young children with zero to 24 months of listening experience.
Total Score on Auditory Skills Checklist (ASC) | Up to 12 Months Post-Activation
  Change from baseline in Total Score on the Auditory Skills Checklist (ASC). Total Score ranges from zero to 70, with higher scores indicating development of increasingly complex listening skills. The Auditory Skills Checklist is intended for children from zero to 18 years of age.
Speech recognition testing in the implanted ear(s) | Up to 12 Month Post-Activation
  Percent change from baseline scores on speech recognition testing with words in quiet and sentences in quiet and noise.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Miami Health System, Miami, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Oregon Health and Sciences University, Portland, Oregon
  - ENT for Children, Coppell, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin